CLINICAL TRIAL: NCT06790368
Title: Prospective Clinical Follow-up to Evaluate the Safety of Immunotherapy for the Treatment of Hymenoptera Venom Allergy in Real-life Conditions.
Brief Title: Immunotherapy for the Treatment of Hymenoptera Venom Allergy in Real-life Conditions.
Acronym: Venox-23
Status: Recruiting | Type: Observational
Sponsor: Inmunotek S.L. (Industry)
Responsible Party: Sponsor
Other Study IDs: ITK-VENOX-2023-01
Record Dates: First submitted 2024-09-16; First posted 2025-01-24 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Allergy, Insect Venom; Allergy Insect Stinging; Insect Sting Allergy
Keywords: Allergy; Immunotherapy; Apis mellifera; Vespula sp; controlled sting
MeSH Terms: conditions — Venom Hypersensitivity; Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood serum to perform immunological study of total IgE, serum tryptase, and specific IgE, IgG4, IgG1.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients allergic to hymenoptera venom: Patients allergic to hymenoptera venom and receive the clinical recommendation to be treated with VENOX inmunotherapy (ATC code: V01AA07)
  Interventions: Biological: VENOX

INTERVENTIONS:
Biological: VENOX — Treatment with allergy vaccine against Vespula spp. (wasp) or Apis mellifera (bee), as per clinical indication.

SUMMARY:
Observational clinical follow-up to evaluate the safety of immunotherapy for the treatment of hymenoptera venom allergy in real-life conditions. It includes the evaluation of controlled and spontaneous stings. This study will be conducted in Spain (multicentric), multicentric and data will be collected prospectively.

DETAILED DESCRIPTION:
Observational, multicentric (Spain), prospective study and data will be collected properly. The total number of participants is expected to be 80. The patients aged equal or more than 14 years old, sentitized to himenoptera venom, not gender differentiation.

ELIGIBILITY:
Inclusion Criteria:

* The study population consisted of allergic participants indicated for treatment with hymenoptera venom immunotherapy (Apis mellifera or Vespula spp.) according to standard clinical practice.
* Participants of both sexes aged 14 years or more.
* Participants who have not received immunotherapy with hymenoptera venom in the previous 5 years.
* Participants who have agreed to take part in the study and sign the informed consent form. In the case of minors, the patient's parent or guardian must also sign.

Exclusion Criteria:

* Pregnant or breastfeeding women.
* Having received immunotherapy with hymenoptera venom during the 5 years prior to the start of the study.
* Participants who do not agree to participate and/or do not sign the informed consent form.
* Participants who do not comply with medical indications or do not cooperate with immunotherapy treatment.

Min Age: 14 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Participants of both gender aged 14 years or more diagnosed of allergy to Apis mellifera and/or Vespula spp. venom, susceptible to receive ITVH according to standard clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-Emergent adverse reactions (safety and tolerability) in participants diagnosed with allergy to hymenoptera venom (Apis mellifera and/or Vespula spp.). | 12 months
  Evaluation of the severity of reactions in relation to subcutaneous immunotherapy following the indications proposed by the World Allergy Organization (WAO).

SECONDARY OUTCOMES:
Evaluation of the effectiveness of treatment with immunotherapy, once the maintenance dose of 100 μg/mL is reached, in participants suffering spontaneous natural stings during the 1-year follow-up. | 12 months
  Registration of allergic reactions, spontaneous natural stings and a controlled sting test in participants sensitised to hymenoptera venom (Apis mellifera and/or Vespula spp.).
Immunological parameters of the participants after 12 months of treatment. | 12 months
  Immunological study: total IgE, specific IgE, IgG4, IgG1 (total extract and molecular components of Vespula spp. and Apis mellifera). The immunological analysis will be performed according to the usual clinical practice of the site and the serum samples will be stored for the complete analysis in the facilities of the sponsor, using the ALEX technique.
SEAIC (Spanish Society of Allergology and Clinical Immunology) Quality of life Questionnaire for people allergic to hymenoptera venom. | 12 months
  The quality of life questionnaire consists of 14 questions, the first nine questions are mandatory. The score for each question is inverse to the order of the answer, i.e. the first answer scores 7 and the seventh 1. The score shall be obtained by adding up all the questions answered and dividing by the total number of questions answered. .The total score goes from 1 to 7, with 1 indicating the worst quality of life and 7 the best.

CONTACTS AND LOCATIONS:
Overall Officials: Arantza Vega Castro, Principal Investigator — Hospital Universitario de Guadalajara
Locations (3):
- Spain (3):
  - Hospital Universitario Fundación Alcorcón, Alcorcón, Madrid
  - Hospital Reina Sofía, Córdoba
  - Hospital Universitario de Guadalajara, Guadalajara

REFERENCES:
- [Background] Krishna MT, Ewan PW, Diwakar L, Durham SR, Frew AJ, Leech SC, Nasser SM; British Society for Allergy and Clinical Immunology. Diagnosis and management of hymenoptera venom allergy: British Society for Allergy and Clinical Immunology (BSACI) guidelines. Clin Exp Allergy. 2011 Sep;41(9):1201-20. doi: 10.1111/j.1365-2222.2011.03788.x. PMID 21848758
- [Background] Ruiz-Leon B, Martinez San Ireneo M, de la Roca F, Arenas L, Alfaya Arias T, Cordobes C, Marques L, Vega A, Moreno-Aguilar C. The Lights and the Shadows of Controlled Sting Challenge With Hymenoptera. J Investig Allergol Clin Immunol. 2022 Oct 11;32(5):357-366. doi: 10.18176/jiaci.0838. Epub 2022 Jun 22. PMID 35735250
- [Background] Alfaya T, Vega A, Dominguez-Noche C, Ruiz B, Marques L, Sanchez-Morillas L. Longitudinal Validation of the Spanish Version of the Health-Related Quality of Life Questionnaire for Hymenoptera Venom Allergy (HRQLHA). J Investig Allergol Clin Immunol. 2015;25(6):426-30. PMID 26817139
- See also: Comite de Alergia a Himenopteros. "Cuestionario de Calidad de Vida en Alérgicos a Himenópteros". — http://www.seaic.org/.